CLINICAL TRIAL: NCT00585026
Title: Randomized Clinical Trial of Bifocal Lenses Versus Computer-specific Progressive Addition Lenses on Symptoms and Performance on a Computer
Brief Title: Randomized Clinical Trial of Bifocal Lenses Versus Computer-specific Progressive Addition Lenses
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left UAB; protocol administratively terminated by UAB IRB.
Sponsor: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Duam
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2009-12

CONDITIONS: Refractive Error; Presbyopia; Asthenopia; Eyeglasses
Keywords: Refractive error; Asthenopia; Presbyopia; Eyeglasses; Productivity; Visual comfort; Ergonomics
MeSH Terms: conditions — Refractive Errors; Presbyopia; Asthenopia

INTERVENTIONS:
Device: D-28 bifocal lenses and frame
Device: Progressive addition computer lenses and frame

SUMMARY:
This is a research study designed to test the utility of D-shaped bifocal lenses and PRIO Computer Lenses for persons using a computer. We hypothesize that lenses specially designed for computer use may allow more comfortable and productive work on a computer.

DETAILED DESCRIPTION:
This is a research study designed to test the utility of D-shaped bifocal lenses and PRIO Computer Lenses for persons using a computer. These are different types of eyeglass lenses and are commonly used when performing computer work. D-shaped bifocal lenses are designed for general purpose use and PRIO Computer Lenses are progressive addition lenses designed for using a computer and are not useful for driving or other tasks requiring clear distance vision. The study will examine how much work a subject completes during a 2-hr visit to the laboratory (productivity) and how a subject feels when working (symptoms). The UAB Department of Optometry sponsors this research study. Interested individuals must be at least 40 years of age and have relatively good vision in each eye when wearing glasses and to do at least 4-hrs of computer work per workday. There are no other restrictions to enter the study.

Participating subjects will be provided one of two different types of lenses and a choice of eyeglass frames. All subjects will be required to use the pair of glasses provided for all computer work for a period of 4 months. During the fourth and eighth weeks of this period, subjects will be required to complete three short surveys over the phone (10 questions) a day for five days (morning, noon and afternoon) on how the glasses affect their work on a computer and how they feel. These surveys should take about 5 minutes or less to complete. During the fifth or sixth week, subjects would be required to visit the laboratory at the School of Optometry to do 2-hours of editing tasks on a computer and complete the same short survey before beginning and after finishing. Participants would be called once a week to confirm that they are wearing the glasses. These calls would last about 2-3 minutes or less.

Upon qualifying for the study, subjects will be randomly (like the flip of a coin) assigned by a computer to receive either the bifocal lenses or the variable focus computer glasses. This will be a single-blind study, which means that neither your doctors completing the survey and the on-site visit will not be informed which type of glasses the subject is using.

The following periodic measurements will be made during the study: visual and upper extremity comfort (surveys) and productivity (editing task). Subjects will be asked to return to the clinic for 1 2-hr visit. At each visit subjects will be asked if they have experienced any undesirable reactions and how they are tolerating the glasses.

ELIGIBILITY:
Inclusion Criteria:

* 40 yrs of age or greater
* 20/40 or better corrected visual acuity in each eye
* 4 hrs or more of computer use per workday

Exclusion Criteria:

* None

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
visual comfort index
productivity (correct words edited per hour)

CONTACTS AND LOCATIONS:
Overall Officials: Kent M. Daum, O.D., Ph.D., Principal Investigator — School of Optometry, University of Alabama at Birmingham
Locations (1):
- School of Optometry, Birmingham, Alabama, United States